## **IRB-Approved Consent Forms for:**

Preventing Sexual Violence Through a Comprehensive Peer-Led Initiative: A Process and Outcome Evaluation

NCT03207386

July 29, 2019

### **Contents:**

Informed consent: Youth Surveys Informed consent: Adult Surveys Informed consent: Youth Photovoice Informed consent: Adult Photovoice

Informed consent: Youth Research Working Group

Informed consent: Youth Focus Group
Informed consent: Adult Focus Group
Informed consent: RPAB youth
Informed consent: RPAB Adult
Informed consent: Key Informant
Informed consent: Youth Interviews

## **Informed Consent: Youth survey**

## IRB #6594

## **Fast Facts**

- ✓ Youth VIP is an exciting project that will allow youth and adults to work together to create programs that we hope will create a safer Rapid City.
- ✓ Surveys are important to see if and how programs are working to keep students safe, healthy, and happy.
- ✓ Students will take 6 short surveys over 3 academic years. This is a one-time form for all of the surveys. If you say "yes" today, you can call or email the Youth VIP research team to take your student out of the study for later surveys.
- ✓ Surveys will be online using computers or smart phones.
- ✓ Your student will NOT put his/her name on the online survey, and researchers will not know who gave what answers to the questions.
- ✓ Students will be asked questions about what they do well, how they help friends stay safe, their role models, and whether they have been hurt by other students.
- ✓ Like school staff, if a student tells a researcher face-to-face that a student is in danger, then the researcher needs to tell someone, like a counselor, who can help.
- ✓ Students will be given information about places in Rapid City that can help students and their friends stay healthy.

### Purpose:

Youth VIP is a program that brings students and adults together to create programs to help students build a healthy future. Learn more at: <a href="www.YouthVIP.org">www.YouthVIP.org</a>. YouthVIP helps students learn skills in order to avoid risky situations. Surveys are a helpful way to give schools and parents information about what students in Rapid City think, and help us see if programs like YouthVIP make student problems happen less and student success happen more.

## **Description of the Study:**

Answer questions on a short 20-minute survey at 6 different times over the next 3 academic years. You can view the survey at <a href="www.YouthVIP.org">www.YouthVIP.org</a>. Surveys will happen in school. Your student will not miss any class assignments. Answer questions about things like their age, what they think about the problems students face, how much they help friends, and whether they have ever had problems like bullying or unwanted sexual experiences from other students. Your student twill also be asked to list names of adults and other students who they look up to so that we can make sure those people are invited to be part of the YouthVIP programs.

### **Voluntary Participation and Right to Withdraw:**

If you do not want your student to do the survey, or your student doesn't want to answer the questions, they can work on something like homework. If you or your student choose not to participate, then your student will not be eligible for the gift card drawings. You can withdraw your student at any time from the project by emailing, calling, or texting us. Your student can stop at any point too. It is completely up to you if you want to let your student take the surveys. If you start by saying "yes" that your student can take the surveys, you can change your mind by calling, texting, or emailing us. After you turn in this form, we will attempt to reach you to confirm that you do or do not want your student to participate.

Even if you say "yes" your student can do the survey, your student will also be asked to choose if he or she wants to answer the questions. As long as your student starts the survey, they can be part of the gift card drawing.

### **Confidentiality:**

The research team plans to keep your student's responses private. Your student's name will not be on the survey. Computer IP addresses are not part of the information we collect even though the survey is done online. Your student does have to be able to take the survey on a computer without any help from anyone else; this is so we can protect the privacy of your student's answers. Your student's name WILL NOT be on any survey questions they answer. A separate researcher will make up numbers to use instead of your student's name on the surveys. That person will never see any answers to survey questions. That person will only put names with ID numbers and the list of those will be destroyed once all surveys are done. Information on these surveys will not become part of school records. No one at the school will see your student's answers. All answers that your child gives to the researchers will be kept private by us, except as described in this paragraph. This study has been given a Certificate of Confidentiality, which means that anything your child tells us will not have to be released to anyone, even if a court orders us to do so, unless you say it's okay. If your student comes up and tells us face-toface, out loud, during the survey about student abuse and/or that they want to hurt themselves or someone else, we will tell others who can make sure your student is safe, just like teachers would do. This is only if they tell us in person, not on the survey. If people have a complaint about the research then the UNH committee that supervises research to make sure that it is being done safely might be able to see some of the survey answers, but your student's name won't be on any of the answers. We will ask for information like your student's address and a working phone number or email to reach him/her if he/she wins the gift card drawing, or send your student a link to the survey if he/she is absent from class when the survey happens. We will keep phone numbers and emails private and separate from survey answers. Your student will get to be in another gift card drawing for filling out the phone/email information. We will also let the person at your student's school who is helping us with this project know if your student missed a survey so that this person can remind your student to take it, if your student wishes to do so. We might also try to call you if your student misses a survey to see if you could remind your student to take the survey.

Information from the surveys will be given back to parents and to schools in short reports that describe the answers of groups of hundreds of students together. Your student's name will never be mentioned in any reports or papers. All data is put together so it is impossible in a report or paper to tell what individual students said on the surveys.

#### **Potential Benefits:**

Most students report that they like being in projects like this because they get to have their voice heard and help others in their community.

### **Potential Risks:**

The survey asks questions including some, like bullying or unwanted sexual experiences (that peers do to one another). We know from a lot of previous research that asking students questions like the ones asked in our survey rarely makes students feel upset or embarrassed. Surveys also do not cause students to do behaviors; for example, asking students about drinking does not make them drink. All students

who take the survey will get information to connect them to someone, like the school counselor, to talk to if they want to.

# **Future Questions and Concerns:**

## **Informed Consent: Adult survey**

## IRB #6594

#### **Fast Facts**

- ✓ Complete one survey in the spring of 2018. We will also contact you again with your permission about a second survey in the spring of 2020.
- ✓ Provide contact information for the gift card drawing (and future survey if you are willing). Your name will not be associated with your survey answers. We will put your contact information for the gift card in a database stored separate from your answers. Your answers will be kept private.
- ✓ After the first survey we will give away six \$50 gift cards. We will give away four \$100 gift cards for the second survey.
- ✓ At the end of the survey you will get information about people in the community you can talk to if you want to learn more.
- ✓ If you tell a researcher face-to-face that a child is in danger then the researcher needs to tell appropriate people such as school staff who can help the child feel safe. This is the same as what school staff do. We will not be asking you questions about this on the survey so you would have to tell us face to face for this to be an issue.
- ✓ The survey is your choice. If you start the survey, you can stop at any time and decide not to take future surveys.

### Purpose:

We want to hear what adults think about how to help youth have happy and healthy futures. We are asking you to do two surveys. One now and one in about 2 years from now.

## **Description of the Study:**

You will be asked questions about things like: what you think youth in Rapid City do well; what challenges they face; how to help youth have healthy relationships; and how parent/guardians, school staff, and adults who work with youth in the community can help youth be happy and healthy.

Adults who take the survey will be entered into a gift card drawing so; we will ask for information like your address and a good phone number or email to reach you so that we can let you know if you win the gift card. We will also send you the link to take a future survey. You do not have to provide your contact information if you do not want to be entered in the gift card drawing. You can also enter the gift card drawing without us contacting you for the future survey, if you just want to complete this survey.

## **Voluntary Participation and Right to Withdraw:**

The survey is your choice. If you start the survey, you can stop at any time and decide not to take future surveys.

## **Confidentiality:**

The research team plans to keep your responses private and report answers as groups of people who took the survey. Computer IP addresses are not part of the information we collect even though the survey is done online. We will work to protect this privacy except as described in this paragraph. This study has been given a Certificate of Confidentiality, which means that anything you tell us on the survey will not have to be released to anyone, even if a court orders us to do so, unless you say it's okay. If you tell us during a survey session about child abuse and/or that you want to hurt yourself or

someone else, we will tell others who can make sure you are safe, but we do not ask specific questions about these things.

### **Potential Benefits:**

You are helping science so that we can learn better ways to help middle and high school students be healthy and have positive futures. A lot of adults say that they like taking surveys like these because they feel like they have a voice about what is going on in their community. The voices of adults are critical to promoting healthy futures for youth.

## **Potential Risks:**

If other individuals (e.g., spouse, children) have access to your computer they might be able to view your web browsing history, including a link to this survey.

Information on how to delete your web browsing history:

http://www.computerhope.com/issues/ch000510.htm

## **Future Questions and Concerns:**

The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email (Katie.Edwards@unh.edu). If you have questions about your rights as a research subject, you may contact Melissa McGee in UNH Research Integrity Services at 603-862-2003 or melissa.mcgee@unh.edu to discuss them.

| ervices at 603-862-2003 or melissa.mcgee@unh.edu to discuss them. |
|---|
| Yes, I am willing to take the survey (please fill out the gift card information below) |
| No, I am not willing to take the survey (Thank you for your time) |

#### **Informed Consent: Photovoice- Youth**

IRB #6594

## **Purpose:**

Youth VIP is a program that brings students and adults together to create programs to help students build a healthy future. Learn more at: www.YouthVIP.orgYouthVIP helps students learn skills in order to avoid risky situations. YouthVIP is about giving students a voice. Photovoice is a type of research that helps people in communities, including youth, show others what they think and feel about their community. They do this by taking photos, discussing photos in a group, and then creating a community event where they show the photos and talk about what they learned from the group. The group will meet 7 times.

## **Description of the Study:**

Your student will get training about things like how to take photos, ethical and safety issues about taking photographs, and how photographs can be a way to express thoughts and feelings about our community.

Each teen will get a digital camera to use, tips on how to use it, and practice using the camera to make sure they are comfortable using it.

At the end of the training session, your teen and the other project participants will decide on the topic they'd like to explore with your cameras. This is called a "photo-assignment." We will also plan a date and time when we will all come back together to discuss the photographs they have taken to complete the first photo-assignment. Before these discussions each teen will look at the photos they have taken, choose one to present to the group, and write some ideas about their photo to bring to the group discussion.

There will be 4 photo discussion sessions, approximately one every two weeks, during the project. During the Photo-discussion Group Sessions (about 1.5 hours each), we (your child, the project staff and the other participants) will all meet together to talk about the photos taken. Your teen will be asked to give their permission to have these "photo-discussions" audio recorded so that we can keep track of the groups' ideas.

Some of these meetings may include Dr. Banyard (one of the main researchers on this project) and Dr. Lightfoot (a national expert in Photovoice with youth) who will use Skype or some other type of remote meeting software to participate in these meetings with youth and the adult supervisor on site in Rapid City.

There will be 2 wrap-up sessions (about 1.5 hours each) where the group will talk about the ideas from all the meetings and plan a community event to talk show the photos and ideas.

### **Voluntary Participation and Right to Withdraw:**

It is completely up to you if you want to let your student do Photovoice.

If you start by saying "yes" that your student can do Photovoice, you can change your mind by calling, texting, or emailing us and having your student return the camera.

Even if you say "yes" your student can do the survey, your student will also be asked to choose if he or she wants to be part of Photovoice.

#### **Confidentiality:**

All answers that your child gives to the researchers will be kept private by us, except as described in this paragraph. This study has been given a Certificate of Confidentiality, which means that anything your child tell us will not have to be released to anyone, even if a court orders us to do so, unless you say it's okay. If your student comes up and tells us face-to-face, out loud, during the photovoice sessions about

student abuse and/or that they want to hurt themselves or someone else, we will tell others who can make sure your student is safe, just like teachers would do. This is only if they tell us in person. Your child's name will not be used during group discussions. We will not use names or personal information on photographs or ideas that are part of exhibits, presentations or publications. Each youth will be asked to create a pseudonym or fake name for the project. Youth will be trained in best practices for taking photos including not taking photographs of faces of people, using photograph consent forms when taking a photo that involves people, and training in photovoice safety. It is possible that other youth in group meetings might talk about what takes place in group discussions of photographs. If people have a complaint about the research then the UNH committee that supervises research to make sure that it is being done safely might be able to see some of the survey answers, but your student's name won't be on any of the answers.

The photographs are taken as part of a project to talk about strengths and concerns of youth in Rapid City related to violence prevention. The photographs will be used to teach the community about what teens think and how youth voices and leadership can help improve violence prevention including the prevention of unhealthy relationships. Your child's photographs will be used to start discussion about community in the group sessions. Some photographs may be included in public exhibits, presentations, or publications. You student should only share and photograph what they consider appropriate and comfortable. With your students' permission, some of their photographs will be used for this project. At the end of the study, your child will receive digital copies of all of the photographs they took. The coinvestigators will keep the photograph files to be used only for educational purposes if your child agrees that they can. Educational purposes may include public exhibits, presentations, and/or reports or future projects. No names are used on photographs that are displayed in exhibits or publications or presentations. Information collected during the meetings and interviews will be stored on password-protected computers, and in files designated for this project. Access will be limited to the researchers. All data stored in computers will have password protection and all paper files will be secured in a locked storage file.

### **Potential Benefits:**

The photographs are taken as part of a project to talk about strengths and concerns of youth in Rapid City related to violence prevention. The photographs will be used to teach the community about what teens think and how youth voices and leadership can help improve violence prevention including the prevention of unhealthy relationships. Your child's photographs will be used to start discussion about community in the group sessions.

#### **Potential Risks:**

It is possible that other youth in group meetings might talk about what takes place in group discussions of photographs.

## **Future Questions and Concerns:**

This project is funded by the National Center for Injury Prevention and Control at the Centers for Disease Control and Prevention. The principal investigator is Dr. Katie Edwards, Associate Professor at the University of New Hampshire (UNH). You can contact Dr. Edwards at the phone or email above. If you have questions about your student's rights as a research subject, you may contact Melissa McGee (UNH Research Integrity Services) at 603-862-2003 or Melissa.mcgee@unh.edu.

| Student Name | _Grade during 2017-2018 |
|-----------------------------------|-------------------------|
| School Attending during 2017-2018 | <u> </u> |

| Legal Guardian Printed Name Legal Guardian Signature |
|---|
| YES, my Student can be part of the Photovoice project or |
| NO, my Student cannot be part of Photovoice |
| (This form is for you as a parent to say YES or NO to your student being part of Photovoice) |
| PLEASE RETURN AS SOON AS POSSIBLE |

#### **Informed Consent: Photovoice-Adult**

IRB #6594

## **Purpose:**

YouthVIP is a program that brings students and adults together to create programs to help students build a healthy future. Learn more at: www.YouthVIP.orgYouthVIP helps students learn skills in order to avoid risky situations. Youth VIP is about giving students a voice. Photovoice is a type of research that helps people in communities show others what they think and feel about their community. They do this by taking photos, discussing photos in a group, and then having a community event where they show the photos and talk about what they learned from the group. The group will meet 7 times plus the community forum. We have a separate Photovoice project for youth. This project is for parents/guardians to learn more about your views about how to help youth be happy and healthy.

## **Description of the Study:**

You will get training about things like how to take photos, ethical and safety issues about taking photographs, and how photographs can be a way to express thoughts and feelings about our community. You will get a digital camera to use, tips on how to use it, and practice using the camera to make sure you are comfortable using it. At the end of the training session, you and the other project participants will decide on the topic you'd like to explore with your cameras. This is called a "photoassignment." We will also plan a date and time when we will all come back together to talk about the photographs they have taken to complete the first photo-assignment. Before these meetings each of you in the group will look at the photos you have taken, choose one to present to the group, and write some ideas about your photo to bring to the group discussion. There will be 4 photo discussion sessions, approximately one every two weeks, during the project. During the Photo-discussion Group Sessions (about 1.5 hours each), we (you, the project staff and the other participants) will all meet together to talk about the photos taken. You are being asked to give your permission to have these "photodiscussions" audio recorded so that we can keep track of the groups' ideas. Some of these meetings may include Dr. Banyard (one of the main researchers on this project) and Dr. Lightfoot (a national expert in Photovoice with youth) who will use Skype or some other type of remote meeting software to participate in these meetings with you and project leaders on site in Rapid City. There will be 2 wrap-up sessions (about 1.5 hours each) where the group will talk about the ideas from all the meetings and plan a community event to talk show the photos and ideas.

### **Voluntary Participation and Right to Withdraw:**

It is completely up to you if you want to do Photovoice. If you start by saying "yes", you can change your mind by calling, texting, or emailing us and returning the camera.

## **Confidentiality:**

Things you say in the photovoice meetings and photos you take will not have your name on them so that we can protect your privacy, except as described in this paragraph. This study has been given a Certificate of Confidentiality, which means that anything you tell us will not have to be released to anyone, even if a court orders us to do so, unless you say it's okay. If you tell us during the photovoice sessions about child abuse and/or that you want to hurt yourself or someone else, we will tell others who can make sure your you are safe, but we do not ask specific questions about these things. Your name will not be used during group discussions. We will not use names or personal information on photographs or quotes or ideas that are part of exhibits, presentations or publications. Each person in the group will be asked to create a pseudonym or fake name for the project. You will learn how to take

photos safely and respecting others including not taking photographs of faces of people, using photograph consent forms when taking a photo that involves people, and training in photovoice safety. It is possible that other people in group meetings might talk about what takes place in group discussions of photographs. If people have a complaint about the research then the UNH committee that supervises research to make sure that it is being done safely might be able to see some of the transcripts of the group discussions and the photos, but your name won't be on the photos or in the transcripts.

#### **Potential Benefits:**

The photographs are taken as part of a project to talk about strengths and concerns of youth in Rapid City related to violence prevention. The photographs will be used to teach the community about what parents/guardians think about how to help youth have a voice and leadership can help improve violence prevention including the prevention of unhealthy relationships. Your photographs will be used to start discussion about community in the group sessions. Some photographs may be included in public exhibits, presentations, or publications. You should only share and photograph what you consider appropriate and comfortable.

#### **Potential Risks:**

You may feel uncomfortable going out to take pictures, but we will talk about this at our meetings. It is possible that you may feel emotional distress or sadness during the discussion, but please keep in mind that you can stop being part of Photovoice, leave the discussion room, or ask the project staff to turn off the audio recorder at any time. You are not required to discuss any issues that make you feel uncomfortable.

#### **Future Questions and Concerns:**

This project is funded by the National Center for Injury Prevention and Control at the Centers for Disease Control and Prevention. The co-principal investigator is Dr. Victoria Banyard, Professor at the University of New Hampshire (UNH). You can contact Dr. Banyard at the phone or email above. If you have questions about your rights as a research subject, you may contact Melissa McGee (UNH Research Integrity Services) at 603-862-2003 or Melissa.mcgee@unh.edu.Vic\_Consent4. Please click one of the options below:

| I agree to be part of the Adult | Photovoice project wit | h Youth VIP. I have | e read and understood the |
|---|---|---|---|
| description of the project on | the following | | |
| pages | | | |
| Yc | urPrinted Name | Your Signature | |

## **Informed Consent: Youth Research Working Group Survey**

IRB #6594

## **Purpose:**

We understand that you are the parent or guardian of a teenager in 6th-12th grade. This teen decided to participate in the Youth Research Working Group (YRWG) which meets once a month to learn about the research process and engage in science. Your teen is invited to participate in a research project focused on gathering information so that we can better understand how the YRWG is working to help youth learn and become engaged in science. The research is being conducted by Dr. Katie Edwards from the University of New Hampshire and research assistants on the Youth VIP project. Please note that if your teen is 18 years of age or older, he or she is legally allowed to make a decision (without parental permission) about participating in this project. Your teen's responses will be combined with responses from a minimum of 5 other people.

## **Description of the Study:**

During a 10-minute time period, your teen will: Complete a survey that asks questions about demographics like age and race. Answer questions about why they decided to join the YRWG, what they are learning, and what they would like to see changed.

## **Voluntary Participation and Right to Withdraw:**

Participation in all parts of this study is up to you and you are free to allow your teen to be part of the research or not. You have the right to take your teen out of the study at any time. Your teen also has the right to quit the study at any time, including the right to stop during the demographic questions and group discussion. There is no penalty or negative consequences for stopping or quitting the study. Your teen also has the right to refuse to answer any questions in the questionnaires or interview.

## Confidentiality:

All answers that your child gives to the researchers will be kept private by us, except as described in this paragraph. This study has been given a Certificate of Confidentiality, which means that anything your child tell us will not have to be released to anyone, even if a court orders us to do so, unless you say it's okay. If your student comes up and tells us face-to-face, out loud, during the YRWG sessions about student abuse and/or that they want to hurt themselves or someone else, we will tell others who can make sure your student is safe, just like teachers would do. Your teen's responses will be reported in terms of groups of participants rather than as individual cases. However, in presentations and publications, participants' responses may be used in the form of quotations, but no names or other identifying information will be included. All of your teen's data will be stored in a locked office in Rapid City, SD before it is transported back to Dr. Edwards' private and locked research laboratory at the University of New Hampshire. Your teen's de-identified data will be transported with other people's de-identified data from the Rapid City, SD office to Dr. Edwards laboratory in Durham, NH through a secure and encrypted server (if electronic data) or through a locked fireproof box that will remain with Dr. Edwards or another member of her team during flight and automobile transportation from Rapid City SD to Durham, NH (if paper data).

#### **Potential Benefits:**

Benefits of your teen's participation include having their voice be heard on what they learned, liked, and would like to change about the Youth Research Working Group. With this information we can optimize

how much the students enjoy and engage in the lessons. People often comment that they enjoy being part of projects like this and being involved in the process of creating a group they can enjoy.

#### **Potential Risks:**

A possible risk includes your teen feeling uncomfortable answering questions about what they are learning or if they want any changes to the program. This discomfort is very unlikely, in fact most people report they benefit by their participation in this type of research. If they feel uncomfortable at any point they can stop taking the survey or skip questions they don't want to answer. Another possible risk is a breach in confidentiality but we have put a lot of protections in place to keep your teen's information private, although there are a few exceptions. However, as we noted above, the exceptions to this are:

1) if your teen tells us (spontaneously) about child abuse or disclosure of an intention to harm self or others, we are required to report to the proper authorities; or 2) there is a rare chance that the University of New Hampshire Institutional Review Board (IRB) will request access to data (e.g., if a participant filed a complaint) (however, in this situation you will not be identified personally).

## **Future Questions and Concerns:**

The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email (Katie.Edwards@unh.edu). If you have questions about your teen's rights as a research subject, you may contact Dr. Julie Simpson in UNH Research Integrity Services at 603-862-2003 or Julie.Simpson@unh.edu to discuss them. I have read and understood the description of the YRWG process evaluation survey. I understand that participation is completely voluntary. \_\_\_\_\_ I agree to have him/her participate in the research project. I DO NOT agree to have him/her participate in the research \_\_\_\_\_Student project.\_\_\_ NameDate Legal Guardian Printed Name Legal Guardian Signature Position with the

Department of Human Services / Juvenile Court, if applicable

## **Informed Consent: Adult Focus Group**

IRB #6594

## Purpose:

The purpose of this study is to collect information about perceptions on why problems like sexual violence, bullying, and dating violence happen among teens in Rapid City, SD and how to prevent these problems in Rapid City, SD. We will ask you to participate in a group discussion with other adults about your ideas for how to keep teens safe, happy, and healthy. We will not be asking you about any personal experiences with interpersonal violence, but rather your ideas on why these things happen and your ideas on how to prevent violence in your school and community. We will also ask you to complete a short demographic survey, to get information like your age and gender. It is typical in research studies to ask this information so that researchers can describe the characteristics of individuals who participated in the project. Your responses will be combined with a minimum of 10 other responses from adults.

## **Description of Study:**

During a 90 to 120 minute time period, you will: ②Complete a demographic survey. Participate in a group discussion to get in-depth information on perceptions about why sexual violence happens and how to prevent sexual violence among teens. Receive a \$25 gift card for being in the group discussion. You will receive the gift card even if you decide not to talk. We will also have drinks and snacks for you. You get the drinks and snacks even if you decide not to talk.

### **Voluntary Participation and Right to Withdraw:**

Participation in all parts of this study is up to you. You have the right to quit the study at any time, including the right to stop during the demographic questions and group discussion. There is no penalty or negative consequences for stopping or quitting the study. You also have the right to refuse to answer any questions in the questionnaires or interview. You will receive the \$25 gift card even if you decide to stop participating in the study.

## Confidentiality:

All answers that you give will be kept private, although there are a few exceptions. One of the exceptions to this is disclosures of child abuse or intent to harm self or others (discussed more below), but we will not ask any questions about this in the survey or group discussion. Your responses will be reported in terms of groups of participants rather than as individual cases. However, in presentations and publications, participants' responses may be used in the form of quotations, but no names or other identifying information will be included. The group discussion will be audio-recorded, and then we will type up what was said in the group discussion (and take out any names and identifying information); the audio recording is destroyed after the interview is typed up.

All of your data will be stored in a locked office in Rapid City, SD before it is transported back to Dr. Edwards' private and locked research laboratory at the University of New Hampshire. Your de-identified data will be transported with other people's de-identified data from the Rapid City, SD office to Dr. Edwards laboratory in Durham, NH through a secure and encrypted server (if electronic data) or through a locked fireproof box that will remain with Dr. Edwards or another member of her team during flight and automobile transportation from Rapid City SD to Durham, NH (if paper data).

#### **Potential Benefits:**

Benefits of participation include the opportunity to contribute to the development of an educational program to prevent sexual violence. People often comment that they enjoy being part of projects like this as they learn about relationships and get to have a voice about prevention happening in their community. We will also ask you what you like most about your community and school, which can help people feel like their voice matters.

#### **Potential Risks:**

The primary risk for you involves dealing with emotional topics like violence. However, we know from previous research that it is very unlikely for people to report being upset by their participation in this type of research. In fact, most people report they benefit from being in research like this project. We will offer resource sheets to all participants and connect them to someone if they wish to talk about the topics further.

Another possible risk is a breach in confidentiality but we have put a lot of protections in place to keep your information private, although there are a few exceptions. However, as we noted above, the exceptions to this are: 1) if you tell us (spontaneously) about child abuse or an intention to harm self or others, we are required to report to the proper authorities; or 2) there is a rare chance that the University of New Hampshire Institutional Review Board (IRB) will request access to data (e.g., if a participant filed a complaint) (however, in this situation you will not be identified personally). We also need to let you know that because you will be talking as part of a group, it is possible that other participants in the group may share what was talked about with others. We will ask all participants not to use the names if they talk about the group.

#### **Future Questions and Concerns:**

The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email(Katie.Edwards@unh.edu). If you have questions about your teen's rights as a research subject, you may contact Dr. Julie Simpson in UNH Research Integrity Services at 603-862-2003 or <a href="mailto:Julie.Simpson@unh.edu">Julie.Simpson@unh.edu</a> to discuss them.

| 1, | _CONSENT/AGREE to participate in this research |
|---------|------------------------------------------------|
| project | <del></del> |

## **Informed Consent: Youth Focus Group**

IRB #6594

## **Purpose:**

The purpose of this study is to collect information about teen's perceptions on why problems like sexual violence, bullying, and dating violence happen in Rapid City, SD and how to prevent these problems in Rapid City, SD. We will ask your teen to participate in a group discussion with other teens about their ideas for how to keep teens safe, happy, and healthy. We will not be asking your teen about any personal experiences with interpersonal violence, but rather their ideas on why these things happen and their ideas on how to prevent violence in their school and community. We will also ask your teen to complete a short demographic survey, to get information like their age and gender. It is typical in research studies to ask this information so that researchers can describe the characteristics of individuals who participated in the project. Your teen's responses will be combined with a minimum of 20 other responses from teens.

## **Description of the Study:**

During a 90 to 120 minute time period, your teen will: Complete a demographic survey. Participate in a group discussion to get in-depth information on teen's perceptions about why sexual violence happens and how to prevent sexual violence. Preceive a \$25 gift card for being in the group discussion. Your teen will receive the gift card even if he or she decides not to talk. We will also have refreshments for teens (e.g., drinks and snacks).

## **Voluntary Participation and Right to Withdraw:**

Participation in all parts of this study is up to you and you are free to allow your teen to be part of the research or not. You have the right to take your teen out of the study at any time. Your teen also has the right to quit the study at any time, including the right to stop during the demographic questions and group discussion. There is no penalty or negative consequences for stopping or quitting the study. Your teen also has the right to refuse to answer any questions in the questionnaires or interview. Your teen will receive the \$25 gift card even if he or she decides to stop participating in the study.

### Confidentiality:

All answers that you child gives will be kept private, although there are a few exceptions. One of the exceptions to this is disclosures of child abuse or intent to harm self or others (more information is provided below), but we do not ask any questions about this in the survey or group discussion. Your teen's responses will be reported in terms of groups of participants rather than as individual cases. In presentations and publications, participants' responses may be used in the form of quotations, but no names or other identifying information will be included. The group discussion will be audio-recorded, and then we will type up what was said in the group discussion (and take out any names and identifying information); the audio recording is destroyed after the interview is typed up. All of your teen's data will be stored in a locked office in Rapid City, SD before it is transported back to Dr. Edwards' private and locked research laboratory at the University of New Hampshire. Your teen's de-identified data will be transported with other people's de-identified data from the Rapid City, SD office to Dr. Edwards laboratory in Durham, NH through a secure and encrypted server (if electronic data) or through a locked fireproof box that will remain with Dr. Edwards or another member of her team during flight and automobile transportation from Rapid City SD to Durham, NH (if paper data).

#### **Potential Benefits:**

Benefits of participation include the opportunity to contribute to the development of an educational program to prevent sexual violence. Teens often comment that they enjoy being part of projects like this as they learn about relationships and get to have a voice about prevention happening in their community. We will also ask teens what they like most about their community and school, which can help teens feel like their voice matters.

#### **Potential Risks:**

The primary risk for your teen involves dealing with emotional topics like violence. However, we know from previous research that it is very unlikely for teens to report being upset by their participation in this type of research. In fact, most teens report they benefit from being in research like this project. We will offer resource sheets to all participants and connect them to someone if they wish to talk about the topics further. A second possible risk is a breach of confidentiality, but as described above we have multiple procedures in place to keep your teen's responses private, although there are a few exceptions. The exceptions to this are: 1) in the case of a spontaneous disclosure of child abuse or disclosure of an intention to harm self or others, we are required to report to the proper authorities; or 2) the possibility on rare occasion that the University of New Hampshire Institutional Review Board (IRB) will request access to data (e.g., if a participant filed a complaint) (however, in the latter case your teen will not be identified personally). It is also important to note that because your teen will be talking as part of a group, it is possible that other teens in the group may share what was talked about with others. We will ask all participating teens not to use the names of other teens if they talk about the group.

### **Future Questions and Concerns:**

The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email(Katie.Edwards@unh.edu). If you have questions about your teen's rights as a research subject, you may contact Dr. Julie Simpson in UNH Research Integrity Services at 603-862-2003 or Julie. Simpson@unh.edu to discuss them.

| I attest that the teen:is in my legal custody in my | y relation to him/her as | |
|---|---|---|
| is in the custody of the Department of Human Se | ervices pursuant to the order of the court | [ |
| agree to have him/her participate in the research proje | ect I DO NOT agree to have him/her | |
| participate in the research project | Adolesce | nt's |
| Name | Legal Guardian Printed | |
| Name | Legal Guardian Signature | |
| <br>Date | Position with Depart | ment |
| of Human Services / Juvenile Court, if applicable | | |

## **Informed Consent: RPAB Adult Survey**

IRB #6594

## **Purpose:**

The purpose of this study is to collect information about people's perceptions about RPAB meetings, what is working and what can be improved, and to collect reflections about your interest in participating in this work and how the RPAB is meeting your own goals. Your responses will be combined with responses from a minimum of 10 other people.

## **Description of the Study:**

During a 7-minutetime period, you will: Complete a demographic survey. Answer 5 short open ended questions about your views of the RPAB so far.

## **Voluntary Participation and Right to Withdraw:**

Participation in all parts of this study is up to you and you are free to be part of the research or not. You also have the right to quit the study at any time, including the right to stop during the survey. There is no penalty or negative consequences for stopping or quitting the study.

## **Confidentiality:**

All answers that you give will be kept private, although there are a few exceptions. We do not ask for your name on the survey. One of the exceptions to this is disclosures of child abuse or intent to harm self or others (discussed more below), but we will not ask any questions about this in the survey or interview. Your responses will be reported in terms of groups of participants rather than as individual cases. However, in presentations and publications, participants' responses may be used in the form of quotations, but no names or other identifying information will be included. All of your data will be stored in a locked office in Rapid City, SD before it is transported back to Dr. Edwards' private and locked research laboratory at the University of New Hampshire. Your de-identified data will be transported with other people's de-identified data from the Rapid City, SD office to Dr. Edwards laboratory in Durham, NH through a secure and encrypted server (if electronic data) or through a locked fireproof box that will remain with Dr. Edwards or another member of her team during flight and automobile transportation from Rapid City SD to Durham, NH (if paper data).

## **Potential Benefits:**

Benefits of participation include the opportunity to contribute to the development of an RPAB and to help us document effective practices for launching these types of community groups. People often comment that they enjoy being part of projects like this as they learn about relationships and get to have a voice about prevention happening in their community.

## **Potential Risks:**

The primary risk for you involves dealing with emotional topics like violence. However, we know from previous research that it is very unlikely for people to report being upset by their participation in this type of research. In fact, most people report they benefit from being in research like this project. Another possible risk is a breach in confidentiality but we have put a lot of protections in place to keep your information private, although there are a few exceptions. However, as we noted above, the exceptions to this are: 1) if you tell us (spontaneously) about child abuse or disclosure of an intention to harm self or others, we are required to report to the proper authorities; or 2) there is a rare chance that

the University of New Hampshire Institutional Review Board (IRB) will request access to data (e.g., if a participant filed a complaint) (however, in this situation you will not be identified personally).

## **Future Questions and Concerns:**

The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email (<a href="mailto:Katie.Edwards@unh.edu">Katie.Edwards@unh.edu</a>). If you have questions about your rights as a research subject, you may contact Dr. Julie Simpson in UNH Research Integrity Services at 603-862-2003 or <a href="mailto:Julie.Simpson@unh.edu">Julie.Simpson@unh.edu</a> to discuss them.

| l, | CONSENT/AGREE to participation | ate in this research |
|---------|--------------------------------|-------------------------|
| project | | Participant's Signature |
| Date | | |

### **Informed Consent: RPAB Youth Survey**

IRB #6594

## **Purpose:**

The purpose of this study is to collect information about people's perceptions about RPAB meetings, what is working and what can be improved, and to collect reflections about your interest in participating in this work and how the RPAB is meeting members' own goals. Your teen's responses will be combined with responses from a minimum of 10other people.

## **Description of the Study:**

During a 7minute time period, your teen will Complete a demographic survey. Answer 5 short open ended questions about their views of the RPAB so far. Questions will ask what your teen feels went well at the meeting and what could be improved. These brief surveys will be given at the end of each monthly RPAB meeting (for a total of 12 per year of the project and a potential of 42 over the course of the research study).

## **Confidentiality:**

All answers that you give will be kept private, although there are a few exceptions. We do not ask for your name on the survey. One of the exceptions to this is disclosures of child abuse or intent to harm self or others (discussed more below), but we will not ask any questions about this in the survey or interview. Your responses will be reported in terms of groups of participants rather than as individual cases. However, in presentations and publications, participants' responses may be used in the form of quotations, but no names or other identifying information will be included. All of your data will be stored in a locked office in Rapid City, SD before it is transported back to Dr. Edwards' private and locked research laboratory at the University of New Hampshire. Your de-identified data will be transported with other people's de-identified data from the Rapid City, SD office to Dr. Edwards laboratory in Durham, NH through a secure and encrypted server (if electronic data) or through a locked fireproof box that will remain with Dr. Edwards or another member of her team during flight and automobile transportation from Rapid City SD to Durham, NH (if paper data).

### **Voluntary Participation and Right to Withdraw:**

Participation in all parts of this study is up to you and you are free to allow your teen to be part of the research or not. You have the right to take your teen out of the study at any time. Your teen also has the right to quit the study at any time, including the right to stop during the demographic questions and group discussion. There is no penalty or negative consequences for stopping or quitting the study. Your teen also has the right to refuse to answer any questions in the questionnaires or interview.

## **Potential Benefits:**

Benefits of participation include the opportunity to contribute to the development of an RPAB and to help us document effective practices for launching these types of community groups. People often comment that they enjoy being part of projects like this as they learn about relationships and get to have a voice about prevention happening in their community.

#### **Potential Risks:**

The primary risk for your teen involves dealing with emotional topics like violence. However, we know from previous research that it is very unlikely for people to report being upset by their participation in this type of research. In fact, most people report they benefit from being in research like this project.

Another possible risk is a breach in confidentiality but we have put a lot of protections in place to keep your information private, although there are a few exceptions. However, as we noted above, the exceptions to this are: 1) if you tell us (spontaneously) about child abuse or disclosure of an intention to harm self or others, we are required to report to the proper authorities; or 2) there is a rare chance that the University of New Hampshire Institutional Review Board (IRB) will request access to data (e.g., if a participant filed a complaint) (however, in this situation you will not be identified personally)..

### **Future Questions and Concerns:**

The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email (<a href="mailto:Katie.Edwards@unh.edu">Katie.Edwards@unh.edu</a>). If you have questions about your teen's rights as a research subject, you may contact Dr. Julie Simpson in UNH Research Integrity Services at 603-862-2003 or <a href="mailto:Julie.Simpson@unh.edu">Julie.Simpson@unh.edu</a> to discuss them.

| | | | | | | • | | | | | |
|------------------|---|----|---|--------|---|----|---|----|----|---|----|
| ^ | | ıt | n | $\sim$ | r | 17 | 2 | T1 | io | n | • |
| $\boldsymbol{H}$ | u | ΙL | | u | | ız | а | u | ıv | ш | ١. |

| I have read and understood the description of the RPAB process evaluation survey. | I understand i | that |
|---|---|---|
| participation is completely voluntary. | | |

| I attest that the teen: is in my lea | gal custody in my relation to him/her as |
|---|---|
| is in the order of the court I agree to have | e custody of the Department of Human Services pursuant to the e him/her participate in the research project I DO NOT e research project |
| | e research project. |
| Adolescent's Name | |
| Legal Guardian Printed Name | |
| Legal Guardian Signature | Date |
| | Position with Department of Human Services |
| / Juvenile Court, if applicable | <u> </u> |

### <u>Informed Consent: Youth Programming Interview Consent</u>

IRB #6594

## **Purpose:**

This interview is part of a larger project being done to help youth and adults work together to create programs that prevent dating violence and sexual assault. Your student attended the Youth Leadership Summer Retreat in July/August 2018 and we would like to learn more about his/her experiences to help improve future retreats and programming. The Youth VIP research project based at the University of New Hampshire is working in partnership with South Dakota Network Against Family Violence and Sexual Assault, Teen-UP, and Working Against Violence, Inc. in Rapid City. Youth VIP is about youth and adults creating projects to make Rapid City safer. The purpose of the interview is to learn about the experiences of the youth who attended retreat so we can work to ensure youth voices are heard in this organization and make improvements for future summer retreats.

#### **FAST FACTS:**

Students will do a 30-60minute interview in-person to tell us about their experiences at the retreat, such as, what you liked and didn't like, including: activities, what you learned, and what you found to be challenging. During the interview your student will be recorded so that we can remember everything that was said, but their name will never be associated with their recording. We will write down everything from the recording and then destroy the recording. Your student will NOT use names, but rather, general terms like "a male student or my friend". It is possible that they might feel a little awkward, sad or embarrassed about some of their experiences, but they have the option not to answer if they don't want to. If a student tells a researcher he or she or someone they know is being hurt, then the researcher needs to tell appropriate people such as school staff who can help the student feel safe. This is the same as what school staff do. Students who do the interview will get a \$25gift card at the end of the interview. Participation in this study is expected to present minimal risk to your student.

## **Description of the Study:**

Answer questions during an in-person interview about their experience at the retreat. Tell researchers what they think about the retreat and if they have any ideas for how to change it to make better next time.

### **Voluntary Participation and Right to Withdraw:**

It is completely up to you if you want to let your student do an interview or not. Even if you say "yes" your student can do the interview, your student will also be asked to choose if he or she wants to answer the questions. As long as your student starts the interview, they will be given the gift card.

## Confidentiality

The research team plans to keep your student's responses private and your student's name will not be on the interview or the notes that the researcher writes. If your student tells us during the interview about student abuse and/or that they want to hurt themselves or someone else, we will tell the appropriate individuals to make sure your student is safe, just like teachers or another school staff would do. Also, sometimes people have a complaint about the research and then the UNH committee that reviews research to make sure that it is being done safely might be able to see some of the notes from the interview.

#### **Potential Benefits:**

You and your student are helping science so that we can learn better ways to help middle and high school students be healthy and have positive futures. Students say that they like being a part of projects like these because they learn about relationships and they feel like they have a voice, or a say, about what is going on in their school and community.

### **Potential Risks:**

It is possible that they might feel a little awkward, sad or embarrassed about some of their experiences, but they have the option not to answer if they don't want to.

## **Future Questions and Concerns:**

More information about the Youth VIP project can be found at www.YouthVIP.orgor by emailing Youth.VIP@unh.edu. The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by phone (603-862-3720) or email (Katie.Edwards@unh.edu).If you have questions about your student's rights as a research subject, you may contact Melissa McGee in UNH Research Integrity Services at 603-862-2005 or melissa.mcgee@unh.edu to discuss them.

## **Informed Consent: Key Informant Interview**

IRB #6594

## **Purpose:**

The purpose of this study is to collect information about people's perceptions on current Youth VIP programming and its' effectiveness at reducing dating violence and sexual assault in Rapid City, SD. We will ask you to participate in an interview to get information about your ideas on current YVIP programming as well as how programming has progressed since summer 2018. We will not be asking you about any personal experiences with sexual violence, but rather your ideas and perceptions on the implementation of YVIP programming. We will also ask you about things like, your role in the community, things that have been challenging, memorable moments, youth engagement, improvements, and impacts. Your responses will be combined with responses from other people.

## **Description of the Study:**

During a 45to 60 minute time period, you will: Participate in an interview to get in depth information on perceptions about the implementation of YVIP programming. Receive a \$25 gift card for being in the interview. You will receive the gift card even if you decide to stop participating.

## **Voluntary Participation and Right to Withdraw:**

Participation in all parts of this study is up to you and you are free to be part of the research or not. You also have the right to quit the study at any time, including the right to stop during the demographic questionnaire and interview. There is no penalty or negative consequences for stopping or quitting the study. You will receive the \$25 gift card even if you decide to stop participating in the study.

### **Confidentiality:**

All answers that you give will be kept private, although there are a few exceptions. One of the exceptions to this is disclosures of child abuse or intent to harm self or others (discussed more below), but we will not ask any questions about this in the survey or interview. Your responses will be reported in terms of groups of participants rather than as individual cases. However, in presentations and publications, participants' responses may be used in the form of quotations, but no names or other identifying information will be included. The interview will be audio-recorded, and then we will type up what was said in the interview (and take out any names and identifying information); the audio recording is destroyed after the interview is typed up. All of your data will be stored in a locked office in Rapid City, SD before it is transported back to Dr. Edwards' private and locked research laboratory at the University of New Hampshire. Your de-identified data will be transported with other people's de-identified data from the Rapid City, SD office to Dr. Edwards laboratory in Durham, NH through a secure and encrypted server (if electronic data) or through a locked fireproof box that will remain with Dr. Edwards or another member of her team during flight and automobile transportation from Rapid City SD to Durham, NH (if paper data).

### **Potential Benefits:**

Benefits of participation include the opportunity to contribute to the development of an educational program to prevent sexual violence. People often comment that they enjoy being part of projects like this as they learn about relationships and get to have a voice about prevention happening in their community.

#### **Potential Risks:**

The primary risk for you involves dealing with emotional topics like violence. However, we know from previous research that it is very unlikely for people to report being upset by their participation in this type of research. In fact, most people report they benefit from being in research like this project. We will offer resource sheets to all participants and connect them to someone if they wish to talk about the topics further. Another possible risk is a breach in confidentiality but we have put a lot of protections in place to keep your information private, although there are a few exceptions. However, as we noted above, the exceptions to this are: 1) if you tell us (spontaneously) about child abuse or disclosure of an intention to harm self or others, we are required to report to the proper authorities; or 2) there is a rare chance that the University of New Hampshire Institutional Review Board (IRB) will request access to data (e.g., if a participant filed a complaint) (however, in this situation you will not be identified personally).

#### **Future Questions and Concerns:**

The University of New Hampshire's Institutional Review Board for the Protection of Human Subjects in Research has approved the use of human subjects in this study. If you have any questions about this research project or would like more information before, during, or after the study, you may contact Dr. Katie Edwards by email at Katie.Edwards@unl.edu. This project is funded by the National Center for Injury Prevention and Control at the Centers for Disease Control and Prevention. The principal investigator is Dr. Katie Edwards, Associate Professor at the University of Nebraska Lincoln. If you have questions about your rights as a research subject, you may contact Melissa McGee in UNH Research Integrity Services at 603-862-2005 or melissa.mcgee@unh.edu to discuss them.

| | 05 or melissa.mcgee@unh.edu to discuss them. | |
|---|---|---|
| integrity services at 003-802-20 | os of <u>menssa.megee@dm.edd</u> to discuss them. | |
| l, | _CONSENT/AGREE to participate in this research project | |
| Print Name | Participant's Signature | Date |